CLINICAL TRIAL: NCT02302300
Title: Interest of the Not Invasive Ventilation Used in Meadow and Post-operative of Cardiac Surgery, in Disease Prevention of the Cardiac and/or Lung Complications at the Patients at Risk.
Brief Title: Interest of the Not Invasive Ventilation Used in Meadow and Post-operative of Cardiac Surgery
Acronym: CAPVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC13.0125
Record Dates: First submitted 2014-07-29; First posted 2014-11-27 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Preventive non-invasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manufacturer STELLAR 150 (Experimental): 5 days of non-invasive ventilation at two levels of pressure from it pre-operative, followed by 5 days in post-operative.
  Interventions: Device: Manufacturer STELLAR 150
- Control Group (No Intervention): Standard preparation

INTERVENTIONS:
Device: Manufacturer STELLAR 150 — 5 days of non-invasive ventilation at two levels of pressure from it pre-operative, followed by 5 days in post-operative.
  Arms: Manufacturer STELLAR 150

SUMMARY:
After cardiac surgery, many complications can arise, in particular at the cardiac and lung level and it is true especially as the patient is with comorbidity. A patient will be considered at risk of a cardiac surgery if risk factors are present in preoperative (obesity, Chronic obstructive pulmonary disease (COPD), etc...). The non-invasive ventilation (NIV)developed these last years in the treatment of acute cardiac insufficiency and the hypercapnic COPD exacerbations; its use is more and more envisaged in cardio-thoracic and abdominal surgery services.

Studies showed that the NIV allowed an improvement of the oxygenation, the lung volumes and a decrease of ventilation work. According to these observations, the preventive NIV could reduce the incidence of appearance of the lung and/or cardiac complications at the patients to risk. we estimate 40 to 50%of cardiac surgery patients at a high risk level and we expect to obtain a benefit with this particular population. If we meet our goal (a significant difference in terms of morbi-mortality with the preventive NIV versus classical care), we expect the systematisation of this procedure to all cardiac surgery high risk patients.

ELIGIBILITY:
Inclusion Criteria:

Every patient of more than 18 years, programmed for a cardiac surgery ( valve replacement, coronary bypass, aortic surgery) in the service of "Chirurgie Cardio-Thoracique et Vasculaire" (CCTV) of the CHRU of Brest

* and obesity (BMI > 30 kg/m2
* and/or COPD (stages 1-2 and 3, classification GOLD)
* and/or restrictive syndrome (CPT 80 %)
* and/or cardiac insufficiency (FEVG 55 %)
* and/or syndrome of obesity-hypoventilation not requiring an equipment
* and/or Syndrome of sleep apnea not requiring an equipment

Exclusion Criteria:

* Patients having a contraindication absolved from the NIV
* Patients carrier of a neuro-muscular disease
* Patients carrier of a syndrome of sleep apnea and/or COPD, and sailed
* Hypercapnic patients (with a limit value of PaCO2 > 55 mm Hg)
* Unaffiliated patients to a social diet of safety
* Patients under guardianship or under guardianship
* Patient who can not follow the NIV program as well as the patients of whom the consent was not collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Appearance of cardio-pulmonary complications in postoperative cardiac surgery | 1 month
  Appearance of cardio-pulmonary complications in postoperative cardiac surgery among the complications listed below:
  * Atelectasis
  * Acute respiratory insufficiency
  * Acute cardiac insufficiency
  * Pneumothorax
  * Arrhythmia
  * Myocardial infarction
  * Cardiac tamponade

SECONDARY OUTCOMES:
Determine postoperative mortality; length of stay in intensive care, length of stay in the service of CCTV | 1 and 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, Pr, Principal Investigator — Département de Médecine Interne et de Pneumologie, CHU BREST
Locations (1):
- CHU Brest, Brest, France

REFERENCES:
- [Derived] Goret M, Pluchon K, Le Mao R, Badra A, Oilleau JF, Morvan Y, Beaumont M, Desanglois G, Guegan M, Barnier A, Gut-Gobert C, Tromeur C, Leroyer C, Choplain JN, Khalifa A, Bezon E, Couturaud F. Impact of Noninvasive Ventilation Before and After Cardiac Surgery for Preventing Cardiac and Pulmonary Complications: A Clinical Randomized Trial. Chest. 2025 Jun;167(6):1727-1736. doi: 10.1016/j.chest.2025.02.010. Epub 2025 Feb 19. PMID 39984118